CLINICAL TRIAL: NCT01040988
Title: The ICD/Device Expectations, Adaptations, and Successes (IDEAS) Study: the Relationship Between Implantable Cardioverter-defibrillators, Pacemakers and Psychiatric Symptoms in a Pediatric Population
Brief Title: The Implantable Cardioverter-defibrillators (ICD)/Device Expectations, Adaptations, and Successes Study
Acronym: IDEAS
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, David DeMaso, Psychiatrist-in-Chief, Chairman, & The Leon Eisenberg Chair in Psychiatry, Boston Children's Hospital; George P. Gardner & Olga E. Monks Professor of Child Psychiatry & Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: X09-04-0195
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression; Anxiety; Post-traumatic Stress Disorder
Keywords: Pacemaker; Implantable cardioverter-defibrillator
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pacemaker: Patients meeting entry criteria with a pacemaker in place.
- ICD: Patients meeting entry criteria with an ICD in place.

SUMMARY:
The introduction of pacemakers and implantable cardioverter-defibrillators (ICDs) has substantially changed the medical and surgical management of patients with cardiac rhythm disease. In the case of patients with ICDs, these devices are programmed to deliver a strong electrical shocks. In adults, multiple studies have suggested that patients at risk of receiving shocks from their device have an increased prevalence of anxiety and depression. Very few studies have looked at this question in children. We propose to evaluate a cohort of patients age 6 to 20 with ICDs, compared to a cohort of patients with pacemakers, assessing each group for the presence of depressive and anxiety disorders, including post-traumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 through 20 at the time of enrollment for patients.
* Age ≥18 for caregiver
* Functioning pacemaker or ICD (explanted or inoperative devices do not qualify)
* Informed consent of parent or guardian as well as assent of study participant

Exclusion Criteria:

* Lack of English language fluency in patient and caregiver
* Hospitalization within 4 weeks of visit
* First implantation of ICD or pacemaker within 6 months of study enrollment

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at participating center with pacemakers and ICDs who fit inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To compare the prevalence of depressive and anxiety disorders (including PTSD) in patients with ICDs or pacemakers using a semi-structured psychiatric interview. | One-time measure at enrollment

SECONDARY OUTCOMES:
We will compare scores on standardized self-assessment tools for subsets of depression and anxiety (including PTSD). | One-time at enrollment
We will compare health-related quality of life between pediatric patients with an ICD and those with a pacemaker. | One-time at enrollment
We will examine caregiver adjustment and family functioning in families of patients with ICDs versus families of patients with pacemakers. | One-time at enrollement
We intend to gather descriptive data on how patients in this age group view their devices. | One-time at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Webster, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] DeMaso DR, Lauretti A, Spieth L, van der Feen JR, Jay KS, Gauvreau K, Walsh EP, Berul CI. Psychosocial factors and quality of life in children and adolescents with implantable cardioverter-defibrillators. Am J Cardiol. 2004 Mar 1;93(5):582-7. doi: 10.1016/j.amjcard.2003.11.022. PMID 14996583
- [Derived] Webster G, Panek KA, Labella M, Taylor GA, Gauvreau K, Cecchin F, Martuscello M, Walsh EP, Berul CI, DeMaso DR. Psychiatric functioning and quality of life in young patients with cardiac rhythm devices. Pediatrics. 2014 Apr;133(4):e964-72. doi: 10.1542/peds.2013-1394. Epub 2014 Mar 24. PMID 24664095